CLINICAL TRIAL: NCT00953550
Title: Rapid Sequence Intubation With Rocuronium-Sugammadex Compared With Succinylcholine
Status: Completed | Phase: Phase 4 | Type: Interventional
Sponsor: Rigshospitalet, Denmark (Other)
Collaborators: TrygFonden, Denmark (Industry)
Responsible Party: Lars Rasmussen, Department of Anesthesia, Center of Head and Orthopedics, Copenhagen University Hospital Rigshospitalet
Allocation: Randomized | Model: Parallel | Masking: Triple | Purpose: Treatment
Other Study IDs: 1B-RSI-SU
Record Dates: First submitted 2009-08-05; First posted 2009-08-06 (Estimated); Last update posted 2011-03-02 (Estimated); Status verified 2010-12

CONDITIONS: Rapid Sequence Intubation
MeSH Terms: interventions — Rocuronium; Sugammadex; Succinylcholine

STUDY DESIGN:
Who Masked: Participant, Investigator, Outcomes Assessor
Oversight: Data Monitoring Committee: Yes

ARMS (2):
- Rocuronium-Sugammadex (Experimental)
  Interventions: Drug: Rocuronium-Sugammadex
- Succinylcholine (Active Comparator)
  Interventions: Drug: Succinylcholine

INTERVENTIONS:
Drug: Rocuronium-Sugammadex — Rocuronium 1,0 mg/kg is administered iv initially. Upon intubation Sugammadex is administered 16 mg/kg iv.
  Other Names: Esmeron; Bridion
  Arms: Rocuronium-Sugammadex
Drug: Succinylcholine — 1 mg/kg
  Other Names: Suxameton; Suxamethon
  Arms: Succinylcholine

SUMMARY:
Rapid sequence intubation is used, when there is an elevated risk of aspiration to the lungs of stomach content. It is typically used in acute settings that require acute surgery or in prehospital settings, but also in specific risk patients requiring elective surgery. The reason for conducting rapid sequence intubation is to minimize the risk of pulmonary aspiration and at the same time achieve a fast induction of anaesthesia and intubation. Rapid sequence intubation is a procedure with a high risk of complications in itself. The time period from induction of anaesthesia to intubation is particularly risky, because the patient is apneic. This study addresses this problem by investigating, how quickly spontaneous respiration can be reestablished after a rapid sequence intubation when using Rocuronium-Sugammadex compared to Succinylcholine. This is a pilot protocol that is intended to establish a sample size for the full protocol.

Study hypothesis: The time from correct tube placement to spontaneous respiration is shorter when using Rocuronium/Sugammadex compared to Succinylcholine.

ELIGIBILITY:
Inclusion Criteria:

* Elective surgical patients with a planned rapid sequence induction of anaesthesia.
* Informed consent.
* Legally competent.
* Be able to understand Danish and be able to read the given information in Danish.
* Females can only participate if they have reached menopause, have had hysterectomy performed, use a coil as birthcontrol, or if they are sterilized.

Exclusion Criteria:

* Presence of kidney disease, defined as S-creatinine >0,200 mmol/L.
* Known lung or heart disease, defined as NYHA-class >2 or CCS-class >2.
* Known allergic reactions to Rocuronium, Suxamethon, Propofol or Sugammadex.
* Contraindications to Suxamethon. Including raised P-potassium (>5,0 mmol/L), untreated glaucoma, neuromuscular disorders or disposition to malignant hyperthermia.
* Body mass index of >35 kg/m2.
* Pregnant.
* Breastfeeding.

Ages: 18 Years to 60 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult
Enrollment: 61 (Actual)
Dates: Start 2009-09; Primary Completion 2011-01 (Actual); Study Completion 2011-02 (Actual)

PRIMARY OUTCOMES:
Time from verified correct tube placement after intubation to spontaneous respiration, defined as respiration frequency of >8/minute, tidal volume >3ml/kg and a saturation of >90% for 30 seconds. | 20 minutes

SECONDARY OUTCOMES:
Duration of action. Measured as the time from administration of the neuromuscular blocking agent to the T1-value in Train-of-Four (TOF) returns to >90% of T1-max. | 20 minutes
Intubation Difficulty Scale (IDS) | 20 minutes
Intubation conditions | 20 minutes
Side effect - Muscle ache. | Postoperative (within 24 hours)
Side effect - Tachycardia (>100 beats per minute). | 20 minutes
Side effect - Bradycardia (<50 beats per minute). | 20 minutes
Side effect - Awareness/recall. Evaluated by modified Brice Questionaire. | Postoperative (within 24 hours)

CONTACTS AND LOCATIONS:
Overall Officials: Martin K Sørensen, MD, Principal Investigator — Rigshospitalet, Denmark
Locations (2):
- Denmark (2):
  - Rigshospitalet, Copenhagen
  - Herlev Hospital, Herlev